CLINICAL TRIAL: NCT03888443
Title: Validation of a Bimanual and Scenarized 3D Motion Analysis Protocol of Upper Limbs in Children With Unilateral Spastic Cerebral Palsy
Brief Title: "Be an Airplane Pilot": A Bimanual 3D Motion Analysis in Children With Unilateral Cerebral Palsy
Acronym: BE-API
Status: Completed | Type: Observational
Sponsor: Rennes University Hospital (Other)
Collaborators: M2S lab (Other); IPSEN, biopharmaceutical group (financial support) (Unknown)
Responsible Party: Sponsor
Other Study IDs: 35RC18_8849_BE-API; 2018-A03290-55 (Other: ANSM (French National Agency for Drugs))
Record Dates: First submitted 2019-03-15; First posted 2019-03-25 (Actual); Last update posted 2019-09-23 (Actual); Status verified 2019-02

CONDITIONS: Unilateral Spastic Cerebral Palsy
Keywords: Unilateral cerebral palsy; three-dimensional movement analysis; upper limb; bimanual task; bimanual performance

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- uCP children: 15 Children aged from 6 to 17 with unilateral spastic Cerebral Palsy and a sufficient level of manipulation will realize the bimanual protocol twice separated from 2 to 4 weeks
  Interventions: Device: Bimanual 3D Motion Analysis " Be-API "
- uCP children with botulinum toxin injections: 5 children aged from 6 to 17 with unilateral spastic Cerebral Palsy and a sufficient level of manipulation will realize the bimanual protocol three times
  Interventions: Device: Bimanual 3D Motion Analysis " Be-API "
- healthy volunteers (TDC children): 20 children aged from 6 to 17 (healthy volunteers) will realize the bimanual protocol once
  Interventions: Device: Bimanual 3D Motion Analysis " Be-API "

INTERVENTIONS:
Device: Bimanual 3D Motion Analysis " Be-API " — Movements will be measured using an optoelectronic system (12 cameras) which captures the displacement of 26 markers placed on the upper limbs and trunk of the child, according to the standards of the International Society of Biomechanics.
  The child is installed on a chair and table height (equipment adapted and approved for pediatrics). A game board is installed in front of the child, with objects to handle, set and placed according to its anthropometry (joystick, steering wheel, buzzer, board, chip).

SUMMARY:
Cerebral Palsy, in particular in its unilateral spastic form (uCP), is the main cause of motor disability in children, with a prevalence of 2/1000 births. These children have upper limb motor impairments that hinder the realization of activities of daily life in bimanual situations. 3D motion analysis (3DMA) is an objective and precise tool, considered as the gold standard for gait analysis. The existing 3DMA protocols consist of movements too standardized, in unimanual situations away from gestures of everyday life, or have not been validated in bimanual situations.

In a preliminary study, a 3DMA bimanual protocol was study. it was composed of 4 tasks integrated into a game scenario to have more spontaneity of movements, similar to those experienced by children in daily life. It allows the exploration of all degrees of freedom of the upper limb. Results showed an excellent acceptability and within day reliability on 20 uCP children and 20 typically developing children (TDC) for funct

DETAILED DESCRIPTION:
This is a prospective study for evaluation of a diagnostic and therapeutic tool.

"Be An Airplane Pilot" 3DMA:

The protocol consists of 5 complementary bimanual tasks that are integrated into a scenario game of "becoming an airplane pilot". It allows the exploration of all degrees of freedom of the UL kinematics of the non-dominant/hemiplegic.

The protocol will take place in a session that corresponds to the driving of an airplane and includes several tasks which consist of 5 repetitions of movements (= 5 cycles).

The kinematics of the trunk (flexion-extension, lateral flexions and rotations), shoulder (elevation, plane of elevation, rotations), elbow (flexion-extension and pronosupination) and wrist (flexion-extension and adduction/abduction) will be explored. The calculated kinematic parameters are the range of motion (ROM) and the maximum angle (MAX) of the degrees of freedom (DoF) of interest.

Group 1: uCP children without botulinum toxin injections

The 3DMA protocol will be performed in two sessions separated from 2-4 weeks to explore the between day reliability in uCP children.

During the first session, this will be associated to physiotherapist and occupational therapist evaluation in order to correlate kinematic parameters to clinical score. During the first session, this will be associated to clinical assessment (muscle strength and tone, pinch, grasp) by a physiotherapist and bimanual performance-based measures (Assisting Hand Assessment (AHA) and Abilhand-kids) by an occupational therapist.

Group 2: uCP children with botulinum toxin injections

Five uCP children will perform the BE-API protocol before and after botulinum toxin injections in the upper limb. This treatment is used for its effect on the local reduction of spasticity after intramuscular injection. It is usually proposed to these children every 6-8 months.

Visit 1 is similar to Group 1 with 3DMA, occupational therapy and physiotherapy.

The second 3DMA will be done during the planned visit for toxin injections (2 to 4 weeks after visit 1) and before treatment administration. Injections of botulinum toxins will be followed by rehabilitation's intensification for 4 weeks (physiotherapy and home exercise) according to the usual care of treated patients.

During Visit 3, 4 to 6 weeks after treatment by botulinum toxin injections, children will have 3D analysis for the third time, with assessment in physiotherapy and occupational therapy, comparable to the Visit 1.

Group 3: healthy volunteers (TDC children)

Their participation in the study will consist of a single visit, during which they will realize the 3DMA protocol only.

Clinical measures

For uCP children, with or without toxin injections, descriptive characteristics such as age, sex, hemiplegic side, as well as Manual Ability Classification System (MACS), Bimanual Fine Motor Function (BFMF) and Modified House Classification will be collected in consultation.

The physiotherapy will do a clinical examination of the upper limbs: passive and active measurement of the range of motion by goniometry, muscle strength, motor selectivity, spasticity, grasp and pinch test, and sensitivity.

The evaluation of the bimanual performance will be carried out by a certified occupational therapist with a validated scale: the Assisting Hand Assessment (AHA) and a questionnaire: the Abiland-Kids (10) which will be filled with the parents

ELIGIBILITY:
Inclusion criteria :

uCP children

* Child aged from 6 to 17,
* With Cerebral Palsy as defined by the SCPE, in unilateral spastic form.
* Sufficient level of manipulation (MACS score from I to III)

TDC children

* Child aged from 6 to 17

Exclusion criteria :

uCP children

* Cognitive deficit altering the comprehension of the instructions or visual disturbances not allowing the visualization of the board game
* Upper limb pain (EVA score> 3),
* Botulinum toxin injections or upper extremity surgery in the 3 months before inclusion
* Contraindication to the use of botulinum toxins and no indications as mentioned in the recommendations HAS 2010

TDC children

* Visual disturbances not allowing the visualization of the board game
* Upper limb pain (EVA score> 3),

Ages: 6 Years to 17 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Study Population: * Children with unilateral spastic Cerebral Palsy and a sufficient level of manipulation followed in Physical Medicine and Rehabilitation in Rennes University Hospital
  * Safe volunteers will be recruited among children of the staff of the Rennes University Hospital (except children unit of Department of Physical Medicine and Rehabilitation) and the M2S laboratory.
Sampling Method: Non-Probability Sample
Enrollment: 40 (Actual)
Dates: Start 2019-02-13 (Actual); Primary Completion 2019-06-26 (Actual); Study Completion 2019-06-26 (Actual)

PRIMARY OUTCOMES:
Primary outcome: Between-day reliability of kinematic parameters (MAX and ROM) will be studied by calculating a between-day Intra-class Correlation Coefficient (ICC) and the Standard Measurement Errors (SEM) from the ICC. | At the end of the participation to the study for each uCP children (2- 4 weeks maximum)
  Two kinematic parameters will be studied: MAX (Maximum angle value) and ROM (Range of Motion) parameters, measured in degrees.
  Outcome measures :
  * Between-day reliability of MAX will be studied by calculating a between-day Intra-class Correlation Coefficient (ICC).
  * Between-day reliability of ROM will be studied by calculating a between-day Intra-class Correlation Coefficient (ICC).
  From ICC, Standard Measurement Errors (SEM) can be calculated. SEM represents from how much degree, it can be considered that the fluctuation is unrelated to chance.

CONTACTS AND LOCATIONS:
Overall Officials: Isabelle bonan, Principal Investigator — Rennes University Hospital
Locations (1):
- Rennes University Hospital, Rennes, France

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Cacioppo M, Lempereur M, Marin A, Rauscent H, Cretual A, Brochard S, Bonan I. Motor patterns of the impaired upper limb in children with unilateral cerebral palsy performing bimanual tasks. Clin Biomech (Bristol). 2022 Jul;97:105710. doi: 10.1016/j.clinbiomech.2022.105710. Epub 2022 Jun 22. PMID 35763887
- [Derived] Cacioppo M, Marin A, Rauscent H, Le Pabic E, Gaillard F, Brochard S, Garlantezec R, Cretual A, Bonan I. A new child-friendly 3D bimanual protocol to assess upper limb movement in children with unilateral cerebral palsy: Development and validation. J Electromyogr Kinesiol. 2020 Dec;55:102481. doi: 10.1016/j.jelekin.2020.102481. Epub 2020 Oct 10. PMID 33091791